CLINICAL TRIAL: NCT03804333
Title: SHort Course Accelerated RadiatiON Therapy (SHARON) in Palliative Treatment of Pelvic Cancer: an Interventional, Randomized, Multicentric Study
Brief Title: Short Course Radiation Therapy in Palliative Treatment of Pelvic Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Alessio Giuseppe Morganti, Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RT 15-04 SHARON PELVIS
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Pelvic Cancer; Radiotherapy; Palliative Care
Keywords: short course radiotherapy; symptomatic pelvic lesions
MeSH Terms: conditions — Pelvic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard treatment (Active Comparator): patients in this group are treated with 3000 cGy in 10 daily fractions
  Interventions: Radiation: standard treatment
- short course treatment (Experimental): patients in this group are treated with 2000 cGy in 4 fractions administered twice a day (at least 6-8 hours interval)
  Interventions: Radiation: short course treatment

INTERVENTIONS:
Radiation: standard treatment — 3000 cGy in 10 daily fractions
  Arms: standard treatment
Radiation: short course treatment — 2000 cGy in 4 fractions administered twice a day
  Arms: short course treatment

SUMMARY:
Aim of the study is to assess efficacy of a short course radiation treatment in patients with symptomatic pelvic malignant lesions

DETAILED DESCRIPTION:
standard treatment for pelvic lesions (300 cGy in 10 daily fractions of 300 cGy each) is compared with experimental treatment (2000 cGy in 4 fractions of 500 cGy twice a day) to demonstrate non-inferiority of this scheme

ELIGIBILITY:
Inclusion Criteria:

* symptomatic pelvic malignant lesions (primary solid tumors or metastases from solid tumor)
* age > 18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-3
* no changes in supportive care in the week before radiotherapy

Exclusion Criteria:

* pregnancy
* previous irradiation of the same region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2017-11-08 (Actual); Primary Completion 2022-11-08 (Estimated); Study Completion 2023-11-08 (Estimated)

PRIMARY OUTCOMES:
efficacy of palliation using the short course scheme compared with the standard scheme: Likert scale | 3 months
  reduction of initial symptoms after radiotherapy, assessed with Likert scale (pain, bleeding, diarrhoea, bowel obstruction, polyuria, urinary obstruction, dysuria, lymphedema, vaginal discharge are evaluated as none-mild-moderate-severe)

SECONDARY OUTCOMES:
acute toxicity in the two treatment groups | 3 months
  incidence of treatment-related acute adverse events in the two arms of the study registered using Cooperative Group Common Toxicity Criteria (RTOG)
late toxicity in the two treatment groups | 12 months
  incidence of treatment-related adverse events in the two arms of the study registered using RTOG/European Organisation for Research and Treatment of Cancer (EORTC) Late Radiation Morbility Scoring Schema
Quality of Life (QoL) assessment in the two groups: EORTC questionnaire C15-PAL | 12 months
  changes in QoL after treatment assessed using EORTC questionnaire C15-PAL (a specific questionnaire from EORTC developed to assess the QoL of palliative cancer care patients)

CONTACTS AND LOCATIONS:
Overall Officials: Alessio G Morganti, MD, Principal Investigator — Radiation Oncology Center, Dept of Experimental, Diagnostic and Speciality Medicine-DIMES, University of Bologna, S.Orsola-Malpighi Hospital
Locations (1):
- Radiation Oncology Center, Department of Experimental, Diagnostic and Speciality Medicine- DIMES, University of Bologna, S.Orsola-Malpighi Hospital, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No